CLINICAL TRIAL: NCT06177574
Title: Study of Bictegravir/Emtricitavine/Tenofovir Alafenamide in HIV-1 Infected naïve Patients Using Test and Treat Stategy Rapid-initiation Model of Care: BIC-NOW Clinical Trial (BIC-NOW)
Acronym: BIC-NOW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Carmen Hidalgo Tenorio (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Carmen Hidalgo Tenorio, Principal Investigator, Medical Director of the Early Stage Clinical Trial Unit-IBS.Granada, University Hospital Virgen de las Nieves
Organization: University Hospital Virgen de las Nieves (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIC-NOW
Record Dates: First submitted 2023-12-07; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: HIV Infections
Keywords: HIV; TEST and TREAT; IMPLEMENTATION
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- study group (Experimental): HIV-1 infected adults, ART-naive subjects, who start BIC/FTC/TAF using test and treat strategy recruited at infectious diseases units from various Spanish public healthcare centers.
  Interventions: Drug: BIC/FTC/TAF

INTERVENTIONS:
Drug: BIC/FTC/TAF — TEST and TREAT strategy: Study group will start the intervention at the first visit with their healthcare provider.

SUMMARY:
The goal of this study is to analyze in treatment-naïve HIV patients the antiviral activity, using a test and treat strategy, in real life of BIC/FTC/TAF. Secondary, this study aims to evaluate outcomes for implementation of the evidence based test and treat strategy.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected adults (>17 y.o.)
2. Antiretroviral-naïve.
3. Be able to comply with protocol requirements and instructions.
4. Subject or the subject's representative capable of giving signed informed consent

Exclusion Criteria:

1. Women who are breastfeeding or plan to become pregnant during the study.
2. Patients who in the investigator's judgment, poses a significant drop out risk or life expectancy inferior to study ending.
3. Patients with anticipated need to change the ART before study ending.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
HIV-1 RNA in plasma (week 24) | 24 week
  copies of HIV RNA -1 in plasma at week 24
HIV-1 RNA in plasma week 48 | 48 week
  copies of HIV RNA -1 in plasma at week 48

SECONDARY OUTCOMES:
Medicaction adherence | 48 week
  proportion of pills taken, self-reported
Retention in care | 48 week
  Subjects completing all study visits
Quality of Life patient reported outcomes EQ-5D | 48 week
  effect of test and treat strategy on health related quality of life and HIV-related symptoms to treatment-naïve HIV patients through PROs EQ-5D (Five dimensions descriptive system of quality of live from EuroQoL)
Quality of Life patient reported outcomes dichotomized HIV-Symptoms Index | 48 week
  effect of test and treat strategy on health related quality of life and HIV-related symptoms to treatment-naïve HIV patients through PROs dichotomized HIV-SI
Feasibility of test and treat strategy | 48 week
  Time to full enrolment of 139 eligible treatment-naïve HIV patients at 22 public healthcare centers in Spain and by physicians using screening data reports
demographics and baseline characteristics | 48 week
  Proportion of subjects by patient subgroup (e.g. by gender, age…) with plasma HIV-1 RNA <50 copies/mL at week 48 using FDA Snapshot algorithm
viral resistance | 48 week
  Incidence of treatment-emergent genotypic or/and phenotypic resistence to any ART
antiviral activity | 48 week
  Time to viral suppression and absolute changes from baseline in lymphocyte count at week 48
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 48 week
  Incidence and severity of adverse events and laboratory abnormalities

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Hospital Universitario Virgen de Las Nieves, Granada, Andalusia
  - H JEREZ, Jerez de la Frontera, Cádiz
  - Hospital Universitario Torrecárdenas, Almería
  - Hospital Universitario Puerto Real, INIBICA,, Cadiz
  - Hospital Campus de la Salud, Granada
  - Complejo Hospitalario de Jaén,, Jaén
  - Hospital Clínico San Carlos, Complutense University, CIBERINFEC ISCIII, Madrid, Spain, Madrid
  - Hu Infanta Leonor, Madrid
  - Hu La Princesa, Madrid
  - Ramon Y Cajal, Madrid
  - Hospital General Universitario Santa Lucía, Murcia
  - Hospital Universitario Virgen de la Arrixaca, IMIB,, Murcia
  - Hospital de Son Llàtzer, Palma de Mallorca
  - Hospital Clínico Universitario de Valencia, Valencia
  - HU la Fé, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sequera-Arquelladas S, Vivancos MJ, Vinuesa D, Collado A, Santos IL, Sorni P, Cabello-Clotet N, Montero M, Font CR, Terron A, Galindo MJ, Martinez O, Ryan P, Omar-Mohamed M, Albendin-Iglesias H, Javier R, Romero A, Vallecillos CG, Calleja MA, Hidalgo-Tenorio C. Impact of bictegravir/emtricitabine/tenofovir alafenamide on health-related quality of life and economic outcomes in HIV care: Substudy of the BIC-NOW clinical trial. PLoS One. 2025 Sep 22;20(9):e0323167. doi: 10.1371/journal.pone.0323167. eCollection 2025. PMID 40982450
- [Derived] Hidalgo-Tenorio C, Sequera S, Vivancos MJ, Vinuesa D, Collado A, Santos IL, Sorni P, Cabello-Clotet N, Montero M, Font CR, Terron A, Galindo MJ, Martinez O, Ryan P, Omar-Mohamed M, Albendin-Iglesias H, Javier R, Ruz MAL, Romero A, Garcia-Vallecillos C. Bictegravir/emtricitabine/tenofovir alafenamide as first-line treatment in naive HIV patients in a rapid-initiation model of care: BIC-NOW clinical trial. Int J Antimicrob Agents. 2024 Jun;63(6):107164. doi: 10.1016/j.ijantimicag.2024.107164. Epub 2024 Apr 2. PMID 38574873